CLINICAL TRIAL: NCT06031207
Title: Translation and Psychometric Properties of the Fatigue Severity Scale in Patients With Fibromyalgia
Status: Completed | Type: Observational
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Other Study IDs: REC-UOL-492-08-2023
Record Dates: First submitted 2023-09-03; First posted 2023-09-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2023-09

CONDITIONS: Fibromyalgia
Keywords: Fatigue Severity Scale; Translation; Psychometric Properties
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study will employ a Cross-Sectional Validation Study design. The study will be conducted at the Department of Physical Therapy, University of Lahore Teaching Hospital, located on Defence Road, Lahore.

The anticipated duration of the study will be 09 months, commencing after the approval of the synopsis.

The sample size will be determined following the Kline Method, resulting in a total of 90 participants.

A Purposive Sampling Technique will be utilized to select the study participants.

DETAILED DESCRIPTION:
Study Type: Cross-Sectional Validation Study Location: Department of Physical Therapy, University of Lahore Teaching Hospital, Defence Road, Lahore Duration: 06 months (post-synopsis approval) Sample Size: 90 participants Sampling Technique: Purposive Sampling Consent and Ethics: Participants will provide written informed consent. Ethics approval will be obtained from the University of Lahore Ethics Committee.

Translation of FSS:

The Fatigue Severity Scale (FSS) will be translated into Urdu for data collection.

Two independent bilingual translators will create reports on translation difficulties and rationale.

These reports will inform a consensus meeting to develop a unified Urdu version, with comments documented.

The unified version will be backtranslated into English by native English-speaking translators unaware of the questionnaire's concept.

Expert Committee:

An expert committee comprising physical therapists, linguists, and a methodologist will review both language versions.

The goal is to ensure semantic, idiomatic, experiential, and conceptual equivalence and reach consensus on the final Urdu version of the FSS.

Patient Involvement:

The final Urdu FSS version will be administered to 20 fibromyalgia patients. These patients will also be interviewed to assess their understanding of questionnaire items.

Participants will receive additional information about fibromyalgia to prevent confusion.

Data Collection:

Data will be collected from 100 fibromyalgia patients using the final Urdu FSS version.

A retest will be conducted after 48 hours.

Additional Assessment:

All 90 participants will complete the Multidimensional Fatigue Inventory (MFI).

ELIGIBILITY:
Inclusion Criteria:

* Both genders with age of 18 years and above
* Diagnosed and referred patients of fibromyalgia according to the American College of Rheumatology (ACR) criteria.
* The ability to provide informed consent and wiling to participate in the study.
* Fluency in the study language (i.e. Urdu in this case).

Exclusion Criteria:

* Any other chronic pain condition that could affect fatigue and sleep.
* Diagnosed sleep disorder (such as sleep apnea or insomnia) that could affect the results.
* History of a psychiatric disorder that could affect the results.
* History of substance abuse.
* Participation in any other study that could affect the results at the time of recruitment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fibromyalgia is a disease characterized by chronic pain, stiffness, and tenderness of muscles, tendons, and joints, without detectable inflammation. Fibromyalgia does not cause body damage or deformity. Fatigue affects 90 percent of patients and sleep disorders are common. Patients diagnosed with fibromyalgia according to the American College of Rheumatology (ACR) criteria will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Fatigue Severity Scale | 1 week
  The Fatigue Severity Scale (FSS) is a self-reported measure of fatigue and sleep disturbance in patients with fibromyalgia. It is a 9-item scale that assesses the severity of fatigue, the impact of fatigue on daily activities, and the degree of sleep disturbance. The FSS is a widely used instrument in research and clinical practice, and has been found to be a valid and reliable measure of fatigue and sleep disturbance in patients with fibromyalgia. The FSS items are rated on a 5-point Likert scale, with responses ranging from "not at all" to "extremely." The total score ranges from 0 to 36, with higher scores indicating greater levels of fatigue and sleep disturbance.
Multidimensional Fatigue Inventory | 1 week
  The Multidimensional Fatigue Inventory (MFI) is a self-report questionnaire designed to assess various dimensions of fatigue experienced by individuals. It is commonly used in research and clinical settings to measure and understand fatigue in different contexts. Respondents answer a series of questions related to each dimension on a Likert-type scale, typically ranging from 1 to 5 or 0 to 4. The scores from each dimension are summed to obtain subscale scores, and a total score is often calculated by summing all subscale scores. Higher scores indicate greater levels of fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Memona Khan, MSPT MSK*, Principal Investigator — University of Lahore; Hafiza Sana Ashraf, MSPT MSK, Study Director — University of Lahore
Locations (1):
- University of Lahore Teaching Hospital, Lahore, Punjab Province, Pakistan